CLINICAL TRIAL: NCT00630851
Title: A Six-month, Multicenter, Double-blind, Parallel, Placebo-controlled Study of the Effect on Global/Behavioural/ADL Functions and Tolerability of Aricept in Patients Wtih Severe Alzheimer's Disease Living in an Assisted Care Facility
Brief Title: A Study of the Efficacy and Safety of Aricept in Patients With Severe Alzheimer's Disease Who Are Living in Skilled Nursing Homes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2501017
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Donepezil (Aricept)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil (Aricept) — Donepezil (Aricept) 5 mg tablet orally once daily for 30 days, followed by 10 mg tablet orally once daily to complete 6 months of treatment
  Arms: 1
Drug: Placebo — Matching placebo tablets orally once daily for 6 months
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Aricept in nursing home patients with severe Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Probable or possible Alzheimer's disease
* Living in skilled nursing home

Exclusion Criteria:

* Other types of dementia or psychiatric or neurologic disorders
* Musculoskeletal disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2002-10; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in modified Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory for Severe Alzheimer's Disease (ADCS-ADL-severe) total score | Month 6
Change from baseline in Severe Impairment Battery (SIB) total score | Month 6

SECONDARY OUTCOMES:
Change from baseline in SIB total score | Month 3
Change from baseline in Neuropsychiatric Inventory (NPI) total score | Months 3 and 6
Change from inclusion in Mini Mental State Examination (MMSE) total score | Month 6
Change from baseline in Clinical Global Impression of Improvement (CGI-I) score | Months 3 and 6
Adverse events and laboratory value changes | Months 3 and 6
Change from baseline in modified ADCS-ADL-severe total score | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- Sweden (49):
  - Pfizer Investigational Site, Fritsla, Sweden
  - Pfizer Investigational Site, Alunda
  - Pfizer Investigational Site, Aneby
  - Pfizer Investigational Site, Avesta
  - Pfizer Investigational Site, Åkersberga
  - Pfizer Investigational Site, Årsta
  - Pfizer Investigational Site, Bengtsfors
  - Pfizer Investigational Site, Bergsjö
  - Pfizer Investigational Site, Boden
  - Pfizer Investigational Site, Borlänge
  - Pfizer Investigational Site, Degerfors
  - Pfizer Investigational Site, Eskilstuna
  - Pfizer Investigational Site, Gislaved
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Gullspång
  - Pfizer Investigational Site, Gustavsberg
  - Pfizer Investigational Site, Hedemora
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Ingelstad
  - Pfizer Investigational Site, Jönköping
  - Pfizer Investigational Site, Kalix
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Katrineholm
  - Pfizer Investigational Site, Kristinehamn
  - Pfizer Investigational Site, Lidköping
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Munkfors
  - Pfizer Investigational Site, Nässjö
  - Pfizer Investigational Site, Oxie
  - Pfizer Investigational Site, Östersund
  - Pfizer Investigational Site, Partille
  - Pfizer Investigational Site, Rättvik
  - Pfizer Investigational Site, Sandviken
  - Pfizer Investigational Site, Särö
  - Pfizer Investigational Site, Sjuntorp
  - Pfizer Investigational Site, Sollebrunn
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Sunne
  - Pfizer Investigational Site, Trollhättan
  - Pfizer Investigational Site, Tullinge
  - Pfizer Investigational Site, Tyreso
  - Pfizer Investigational Site, Umeå
  - Pfizer Investigational Site, Upplands Vasby
  - Pfizer Investigational Site, Uppsala
  - Pfizer Investigational Site, Vaxjo
  - Pfizer Investigational Site, Vännäs
  - Pfizer Investigational Site, Värnamo
  - Pfizer Investigational Site, Västerås
  - Pfizer Investigational Site, Visby
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2501017&StudyName=A%20study%20of%20the%20efficacy%20and%20safety%20of%20Aricept%20in%20patients%20with%20severe%20Alzheimer%27s%20disease%20who%20are%20living%20in%20skilled%20nursing%20homes